CLINICAL TRIAL: NCT07378748
Title: Effect of Bedtime Meditation on Spiritual Well-Being and Anxiety in Hemodialysis Patients
Brief Title: Effect of Bedtime Mindfulness Meditation on Anxiety and Spiritual Well-Being in Hemodialysis Patients
Acronym: BM-BOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Wara Gati Murwani, Ners., Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-BMBOM
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Anxiety; Spiritual Well-being
Keywords: Bedtime Meditation; Spiritual Well-Being; Hemodialysis Patients; Anxiety Reduction; BM-BOM
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two parallel groups: an intervention group receiving Bedtime Meditation Based on Mindfulness (BM-BOM) and a control group receiving passive rest without guided mindfulness. Outcomes were measured at baseline and after four weeks of intervention.
Who Masked: Participant
Masking Description: This study used a single-blind design in which participants were blinded to their group allocation. Outcome assessment was conducted using self-reported questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BM-BOM Intervention Group (Experimental): Participants received a 2.5-hour face-to-face mindfulness training delivered by a certified practitioner, followed by guided Bedtime Meditation Based on Mindfulness (BM-BOM) practice during hemodialysis sessions twice weekly for four consecutive weeks. Each session lasted approximately 15 minutes and was delivered using standardized audio guidance consisting of breathing awareness, body scan, and closing reflection.
  Interventions: Behavioral: Bedtime Meditation Based on Mindfulness (BM-BOM)
- Control Group (Passive Rest) (Active Comparator): Participants rested quietly with their eyes closed for approximately 15 minutes at the beginning of each hemodialysis session twice weekly for four weeks, without structured mindfulness guidance. This controlled for time, attention, and treatment environment
  Interventions: Behavioral: Passive Rest (Control)

INTERVENTIONS:
Behavioral: Bedtime Meditation Based on Mindfulness (BM-BOM) — A structured mindfulness-based intervention consisting of guided breathing awareness, body scan, and closing reflection delivered via standardized audio recordings. Participants practiced BM-BOM for approximately 15 minutes during hemodialysis sessions twice per week for four weeks after completing a 2.5-hour introductory training session led by a certified mindfulness practitioner.
  Arms: BM-BOM Intervention Group
Behavioral: Passive Rest (Control) — Participants rested quietly with eyes closed for approximately 15 minutes during hemodialysis sessions without any guided mindfulness or structured intervention.
  Arms: Control Group (Passive Rest)

SUMMARY:
This study evaluates whether Bedtime Meditation Based on Mindfulness (BM-BOM) can reduce anxiety and improve spiritual well-being in patients undergoing hemodialysis.

People receiving long-term hemodialysis often experience emotional stress, anxiety, and spiritual distress due to chronic illness, treatment burden, and lifestyle limitations. These problems may affect their quality of life and overall well-being. Mindfulness meditation is a simple, low-cost, and safe non-drug approach that may help patients feel calmer, more focused, and more spiritually connected.

In this study, adult hemodialysis patients are randomly assigned to one of two groups. The intervention group receives a guided mindfulness meditation program. Participants attend a single 2.5-hour training session led by a certified mindfulness instructor and then practice guided meditation during their hemodialysis sessions twice a week for four weeks using audio recordings. Each session lasts approximately 15 minutes and includes breathing awareness, body awareness, and short reflection.

The control group follows the same schedule and duration but rests quietly with eyes closed without guided meditation.

Participants complete questionnaires before and after the four-week program to measure anxiety and spiritual well-being. The results of this study will help determine whether guided mindfulness meditation can be used as a practical and supportive complementary therapy for patients receiving hemodialysis.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of Bedtime Meditation Based on Mindfulness (BM-BOM) in reducing anxiety and improving spiritual well-being among patients undergoing maintenance hemodialysis.

Hemodialysis patients frequently experience psychological distress, including anxiety, emotional burden, and spiritual challenges associated with long-term treatment dependency, physical limitations, and uncertainty about health outcomes. Although standard hemodialysis care focuses primarily on physiological management, psychosocial and spiritual needs are often insufficiently addressed. Mindfulness-based interventions offer a structured, non-pharmacological approach that promotes present-moment awareness, emotional regulation, relaxation, and adaptive coping. However, evidence regarding their combined effects on anxiety and spiritual well-being in hemodialysis populations remains limited.

This study employs a single-blind randomized controlled design with pre- and post-intervention measurements. Eligible participants are adult patients with stage V chronic kidney disease who have been receiving outpatient hemodialysis for at least three months and are able to communicate effectively and provide informed consent. Participants with severe cognitive impairment, diagnosed psychological disorders, or medical conditions that prevent participation in the intervention are excluded.

A total of 58 participants are randomly allocated in a 1:1 ratio to either the intervention group or the control group using a computer-generated randomization sequence. Participants are blinded to group allocation. Outcomes are assessed using self-reported standardized questionnaires administered at baseline and again after completion of the four-week intervention period.

Participants in the intervention group receive a structured mindfulness program. The program begins with a single 2.5-hour face-to-face training session delivered by a certified mindfulness practitioner, introducing core principles of mindfulness, breathing awareness, and body awareness. Following the training, participants practice guided BM-BOM at the beginning of each hemodialysis session, twice weekly for four consecutive weeks. Each session lasts approximately 15 minutes and is delivered using standardized audio guidance in the Indonesian language. The audio guidance includes three sequential components: focused breathing awareness (approximately 5 minutes), body scan and bodily awareness (approximately 7 minutes), and closing reflection and grounding (approximately 3 minutes). Attendance and adherence are monitored during each session.

Participants in the control group follow the same schedule, setting, and duration but do not receive mindfulness guidance. They are instructed to rest quietly with eyes closed during the first 15 minutes of hemodialysis. This approach controls for time, attention, and environmental exposure while minimizing expectancy effects.

The primary outcomes are changes in spiritual well-being and anxiety levels from baseline to post-intervention. Spiritual well-being is measured using the Indonesian version of the Spiritual Well-Being Scale (SWBS), and anxiety is assessed using the Indonesian version of the Zung Self-Rating Anxiety Scale (ZSARS). Both instruments have demonstrated acceptable validity and reliability in Indonesian populations.

Data analysis includes descriptive statistics to summarize participant characteristics and inferential testing to compare within-group and between-group changes. Normality and homogeneity assumptions are evaluated prior to hypothesis testing. Paired statistical tests are used to assess pre- and post-intervention changes within groups, and independent statistical tests are used to compare outcome differences between groups. Effect sizes are calculated to support interpretation of clinical relevance.

Ethical approval is obtained from the institutional research ethics committee, and all participants provide written informed consent prior to participation. Participant confidentiality is maintained throughout the study in accordance with ethical guidelines.

The findings of this trial aim to provide evidence on the feasibility, safety, and effectiveness of guided mindfulness meditation as a complementary intervention that can be integrated into routine hemodialysis care to support psychological and spiritual well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic kidney disease (CKD) stage V.
* Undergoing outpatient hemodialysis for at least three months.
* Aged 18 years or older.
* Able to communicate effectively.
* Willing to participate and provide written informed consent.

Exclusion Criteria:

* Severe cognitive impairment.
* Diagnosed psychological or psychiatric disorders.
* Any medical condition that prevents participation in the mindfulness intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Spiritual Well-Being Score | Baseline (Week 0) and after 4 weeks of intervention (Week 4)
  Spiritual well-being will be measured using the Indonesian version of the Spiritual Well-Being Scale (SWBS). The SWBS assesses overall spiritual well-being through self-reported questionnaire items. Higher scores indicate better spiritual well-being. The primary outcome is the change in SWBS total score from baseline to post-intervention.

SECONDARY OUTCOMES:
Change in Anxiety Score | Baseline (Week 0) and after 4 weeks of intervention (Week 4)
  Anxiety will be assessed using the Indonesian version of the Zung Self-Rating Anxiety Scale (ZSARS), a 20-item self-reported questionnaire. Higher scores indicate higher anxiety levels. The secondary outcome is the change in ZSARS total score from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- UNS Hospital, Surakarta, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with external researchers. The dataset will remain confidential and will only be accessible to the research team, in accordance with ethical approval and data protection regulations.

REFERENCES:
- [Background] Murwani WG, Rosyid FN, Hudiyawati D. Effect of Bedtime Meditation on Spiritual Well-Being and Anxiety in Hemodialysis Patients: A Randomized Controlled Trial. Manuscript in preparation / submitted for publication, 2025.